CLINICAL TRIAL: NCT02341820
Title: PICTURE Breast L: Patient Information Combined for Local Therapy oUtcome Assessment in bREast Cancer - Longitudinal
Acronym: PICTURE L
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: 8713
Record Dates: First submitted 2015-01-13; First posted 2015-01-19 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2016-10

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; breast conserving surgery; cosmesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This project which is fully funded by the European Union FP7 Program is designed to pull together all the information we obtain from scans and x-rays to design a personalised 3-D digital model of each patient, their anatomy and disease. We can then use this as follows: as (i) an aid to surgical planning to enable objective clinical decision making (ii) a decision support tool to communicate the available treatment options to the patient and facilitate shared decision making and provision of personalised care and (iii) to enable standardised objective evaluation of the aesthetic outcome of the treatment procedures. This study aims to demonstrate the ability of the Virtual Physiological Human concept to empower breast cancer patients and assess the impact on their care and quality of life.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer to affect women in Europe, having a lifetime risk of 1 in 9. It is an increasingly treatable disease, and 10-year survival now exceeds 80%. The primary treatment for breast cancer is surgery, which may be used in conjunction with adjuvant therapies, such as chemotherapy and radiotherapy. Given the high breast cancer survival rate, many women will live for many years with the potentially disfiguring aesthetic consequences of their surgical and therapeutic treatment. A good aesthetic outcome is an important endpoint for breast cancer treatment and is closely related to psychosocial recovery and quality of life.

When a woman faces a breast cancer diagnosis, and surgery is proposed, several options are available. The decision as to which type of surgery to offer patients is largely subjective and based almost exclusively on the judgment and experience of the clinician. The cosmetic outcome of surgery is a function of many factors including tumour size and location, the volume of the breast, its density, and the dose and distribution of radiotherapy. In breast-conserving surgery, there is evidence that approximately 30% of women receive a suboptimal or poor aesthetic outcome; however there is currently no standardised method of identifying these women.

The PICTURE project aims to address these issues by providing objective tools, tailored to the individual patient, to predict the aesthetic outcome of local treatment. Using a combination of 3D photography and routinely acquired radiological images (i.e. mammography, ultrasound and MRI, when available), together with information about the tumour (size, location, shape etc.) we will develop techniques to biomechanically model the anatomy of the breast and the effect of surgical removal of cancerous tissue. This digital patient representation and associated predictive tools will enable alternative surgical strategies to be explored and the consequences of the available options, with respect to the appearance of the breast, to be visualised. This will aid communication with the patient of the type of breast surgery recommended by the surgeon, and will empower patients to take an active role in a shared decision making process.

The study will develop tools to enable the patient's aesthetic appearance after treatment to be objectively evaluated. Current techniques use subjective methods, such as assessment by an expert panel, or computer analysis of 2-dimensional photography to estimate, for instance, breast asymmetry. By adopting recent developments in low cost 3D photography and depth sensing technology, we will develop a standardised, reproducible analysis tool which will base the aesthetic outcome evaluation on both the 3-dimensional shape of the reconstructed breast and its volume. This will establish standardised quality assurance and evaluation procedures, enabling institutions across Europe to be compared and factors that have a positive or negative impact on surgical outcome identified.

In summary, the demonstrator created by the PICTURE project will integrate models of surgical techniques and treatment schemes, clinical patient data, multi-modal imaging and individualised models of patient anatomy to build a personalised, digital representation of the patient. The aim is for this to be used as an aid to surgical planning, via simulation of the cosmetic effects of breast conserving surgery, as a decision support tool to communicate the available options to the patient and to enable standardised evaluation and a safe outcome of the procedure. The demonstrator aims to empower patients and will have a direct impact on their care and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing breast conserving surgery for early breast cancer.
* Willing and able to return for a one-year visit.
* Written informed consent obtained.

Exclusion Criteria:

* Unable to provide written informed consent.
* Younger than 18 years.
* Benign breast disease.
* Women undergoing mastectomy.
* Unable to have an MRI scan (e.g. claustrophobia, too large, etc.).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who are scheduled to undergo breast conserving surgery for early breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Creation of a reliable demonstrator. | One year
  The primary objective of the study is to create a reliable demonstrator (software) by integrating models of surgical techniques and treatment schemes, clinical patient data, multi-modal imaging and individualised models of patient anatomy. The demonstrator will be used as an aid to objective surgical planning, via simulation of the cosmetic effects of breast conserving surgery, as a decision support tool to communicate the available options to the patient and to enable standardised evaluation of the procedure.

SECONDARY OUTCOMES:
Assess health-related quality of life. | One year
  The secondary objective is to assess the health-related quality of life at baseline (before surgery) and one year after surgery, in the women who are participating in this study. Together with characteristics of the patient and the breast tumour, these data will describe the patient group on whom the demonstrator is constructed, which will be used to inform the design and size of a subsequent evaluation study.

CONTACTS AND LOCATIONS:
Overall Officials: Mo Keshtgar, Principal Investigator — Royal Free London
Locations (3):
- Leiden University Medical Center (LUMC), Leiden, Netherlands
- Champalimaud Cancer Center, Lisbon, Portugal
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All requests for data sharing will adhere to the UCL Surgical & Interventional Trials Unit (SITU) data sharing agreement policy. UCL Medical School is supportive of data sharing and will endeavour to assist in requests for data sharing. These data will be held at UCL on secure servers and will not be released to any third parties until the final study report has been published. All requests for access to the data will be formally requested through the use of a SITU data request form which will state the purpose, analysis and publication plans together with the named collaborators. All requests are dealt with on a case by case basis. All requests will be logged and those successful will have a data transfer agreement which will specify appropriate acknowledgement of the Royal Free Hospital, the sponsor, and funders.

REFERENCES:
- See also: EU FP7 website — http://cordis.europa.eu/project/rcn/106628_en.html